CLINICAL TRIAL: NCT00494156
Title: Anticoagulation in the Management of Grade I-III Blunt Cerebrovascular Injuries
Brief Title: Anticoagulation in Blunt Cerebrovascular Injuries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely prior to enrollment of first participant.
Sponsor: C. Clay Cothren, MD (Other)
Responsible Party: Sponsor-Investigator, C. Clay Cothren, MD, Principal Investigator, Denver Health and Hospital Authority
Organization: Denver Health and Hospital Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMIRB 00-508
Record Dates: First submitted 2007-06-25; First posted 2007-06-29 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Carotid Artery Injury; Vertebral Artery Injury
MeSH Terms: conditions — Carotid Artery Injuries | interventions — Heparin; Aspirin; Clopidogrel

INTERVENTIONS:
Drug: heparin
Drug: aspirin and clopidogrel

SUMMARY:
Originally thought to be a rare occurrence, BCVI are now diagnosed in approximately 1% of blunt trauma patients. Initially BCVI were thought to have unavoidable devastating neurologic outcomes. But early reports suggested anticoagulation might decrease these events. If untreated, carotid artery injuries (CAI) have a stoke rate up to 50% depending on injury grade, with increasing stroke rates correlating with increasing grades of injury. Current studies report early treatment with antithrombotics - either heparin or anti-platelet agents - in patients with BCVI markedly reduces stroke rates and resultant neurologic morbidity. As reports of bleeding complications have altered heparin protocols in these patients, the use of antiplatelet agents is attractive. Although heparin has been has been proposed as the gold standard treatment due to its initial empiric use, no comparative studies of antithrombotic agents has been performed.

In sum, Grade I-III blunt carotid and vertebral arterial injuries (BCVI) have the potential for stroke, and should be treated. Heparin has not been shown to clearly improve healing rates compared with antiplatelet therapy. The purpose of this study is to determine whether systemic anticoagulation alters the course of Grade I-III BCVI compared with antiplatelet therapy. The investigators study hypothesis is that Grade I-III BCVI will heal or progress to pseudoaneurysm formation, independent of systemic antithrombotic regimen, and that the combination of aspirin and clopidogrel is equally efficacious in preventing neurologic symptoms compared to systemic heparin associated with Grade I-III BCVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years old with documented grade I-III blunt cerebrovascular injuries.

Exclusion Criteria:

* Pregnancy
* Nasal polyps
* Previous gastrointestinal bleeding secondary to antiplatelet medications
* Contraindication to systemic anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-07; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Neurologic sequelae | during hospital visit

CONTACTS AND LOCATIONS:
Overall Officials: Clay Cothren, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States